CLINICAL TRIAL: NCT02305940
Title: A Phase III Double-blind, Randomised, Placebo Controlled Trial of Long Term Therapy on Exacerbation Rate in Patients With Stable COPD Using Doxycycline
Brief Title: Effects of Long Term Antibiotic Therapy on Exacerbation Rate in Stable COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14IC2030
Record Dates: First submitted 2014-11-20; First posted 2014-12-03 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): Doxycycline: oral dose of 100 mg once daily, for a total duration of 52 weeks.
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Placebo: an oral dose of one capsule once daily, for a total duration of 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — An oral dose of 100 mg of Doxycycline once daily, for a total duration of 52 weeks.
  Arms: Doxycycline
Drug: Placebo — An oral dose of one capsule of placebo once daily, for a total duration of 52 weeks
  Arms: Placebo

SUMMARY:
This study investigates if long term use of the antibiotic doxycycline can reduce exacerbations in COPD patients. Half of the patients will receive doxycycline which the other half will receive a placebo.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common disease which can place a considerable burden on people who suffer from it. COPD exacerbations (periods when symptoms flare up) are a major cause of hospital admission in the UK. Bacterial infections play an important role in the development of COPD and so one possible treatment for COPD is with antibiotics. However, there is little information available about the use of long term antibiotics in the treatment of this disease.

Therefore, the purpose of this study is to investigate if long term use of the antibiotic Doxycycline can reduce exacerbations and improve the outlook for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given
* Confirmed COPD diagnosis
* Severity of disease: Patients with a measured FEV1<80% of predicted normal values.
* At least one treated exacerbation (Patient recalls an episode of symptomatic worsening which was treated and was consistent with a COPD exacerbation) in the previous year.
* Age: ≥ 45 years of age at screening.
* Able to complete questionnaires for health status and symptoms and considered able to comply with the dosing regimen.
* Patients willing to report exacerbations and attend for study visits.

Exclusion Criteria:

* Patients with a known diagnosis of active TB or other chronic respiratory disease in the judgement of the study doctor.
* Hepatic or renal impairment as defined as LFTs > 5XULN, and eGFR<30 ml/min/1.73m2.
* Patients with known hypersensitivity to Tetracyclines, the IMP and/or Placebo including their excipients.
* Patients taking ongoing antibiotic therapy for COPD or other conditions.
* Patients with uncontrolled clinically significant hypertension
* Female patients who are pregnant or planning on becoming pregnant during the study, or are breastfeeding.
* Patients with uncontrolled clinically relevant bradycardia, cardiac arrhythmias or cardiac insufficiency.
* Clinically relevant abnormal electrolyes (sodium or potassium), renal function (urea and creatinine) or liver function (ALT, AST, ALP) that could interfere with the objectives of the trial or safety of the volunteer.
* Patient taking clinically significant contraindicated medication, as per the SmPC for Doxycycline.
* Use of another experimental investigational medicinal product within 3 months of study enrolment. If the IMP used was as part of the NIHR WP2 study then entry to WP3 after a 6 week washout period is permissible.
* Patients with any other condition precluding enrolment in the trial, according to the assessment of the study doctor. This will be documented at screening

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Rate of exacerbations (per person/year) recorded from date of drug issue until date of end of treatment visit. | 12 months

SECONDARY OUTCOMES:
Lung function (spirometry) (FEV1, FVC, FEV1/FVC ratio, FEV1 as % Predicted). | 12 months of treatment
Total and individual component (symptoms, activity, impact) SGRQ scores will be used to measure health status. | 12 months of treatment
Respiratory health status across groups as measured from total number of symptoms in a day and prevalence of individual symptoms recorded on daily diary cards. | 12 months of treatment
Airway bacteria numbers taken from a sputum sample, provided by a subset of patients, at months 3, 6, 9, 12 after drug issue. | 12 months of treatment
Changes in C-reactive protein (CRP) levels from baseline. | 12 months of treatment
Hospital admissions. This data will be collected from Hospital Episode Statistics (HES). | 12 months of treatment
Time to 1st exacerbation measured by diary cards in both therapy and placebo groups. | 12 months of treatment
Rate of exacerbations treated with steroids and antibiotics. | 12 months of treatment
Adherence as measured using pill counts. | 12 months of treatment
Antibiotic resistance measured in the subset of patients (able to produce sputum) from sputum based on standard NHS procedures (not resistant, intermediate, severe, resistant). | 12 months of treatment

OTHER OUTCOMES:
Pre-specified Exploratory Subgroup Analysis | 12 months of treatment
  As co-morbidities for COPD are heterogeneous, exploratory analysis will be carried out to investigate whether there is an interaction with treatment- i.e. to investigate whether outcomes of treatment are either influenced by and/or restricted to patients with particular known co morbidities. The following will be looked at in this study:
  Cardiovascular disease. This included patients receiving treatment for Ischemic Heart Disease, hypertension and heart failure.
  Diabetes and/or known impaired glucose intolerance Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Wisia Wedzicha, MD, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - St Georges University Hospitals NHS Foundation Trust, London
  - Royal Brompton and Harefield Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allinson JP, Vlies BH, Brill SE, Law M, Burnside G, Finney LJ, Alves-Moreira L, Donaldson GC, Calverley PMA, Walker PP, Wedzicha JA. A Double-Blind, Randomized, Placebo-controlled Trial of Long-Term Doxycycline Therapy on Exacerbation Rate in Patients with Stable Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Sep 1;208(5):549-558. doi: 10.1164/rccm.202212-2287OC. PMID 37450935